CLINICAL TRIAL: NCT06513741
Title: Building Stronger Foundations: Exploring a Collaborative Faculty Mentoring Workshop for In-depth Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-6127-17832
Record Dates: First submitted 2024-07-01; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Behavior
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Workshop Participants (Experimental): Educate faculty members to develop personal development plans for becoming effective mentors and mentees
  Interventions: Behavioral: Mentoring Workshop

INTERVENTIONS:
Behavioral: Mentoring Workshop — Faculty mentoring workshop with the title "Faculty Mentoring; building stronger by digging deeper" was designed as a two-day workshop of three hours each for the faculty members of the two institutions at separate times

SUMMARY:
Mentorship training programs demand a paradigm shift from theory-driven approach to hands-on practical approach. This requires prioritisation of preparation of mentors and mentees for their roles through self-awareness and targeted professional development. There is a lack of evidence form health professions education institutions of global south, regarding effectiveness of the workshops in fostering mentorship culture. A mixed method study with convergent parallel design is conducted through a collaborative mentoring workshop; "Faculty Mentoring-Building stronger by digging deeper" by Aga khan University Medical College, Karachi and University of Lahore, Punjab, Pakistan. Objective of the research is to emphasise the importance of faculty mentoring program, roles and responsibilities of mentors and mentees and collecting perceptions of the participants regarding the associated role of institutions. It aims to educate faculty members to develop personal development plans for becoming effective mentors and mentees. The designed intervention is a 12 hour workshop spanned over two days of six hours each with the focus on determining perception of the Medical faculty of two institutions regarding the importance and preparedness of faculty development programs and the focus on self through personal swot translating into a personal development plan. The demographic data of participants was collected before the workshop, during the workshop, and after workshop. Comparison between quantitative findings was done through ANOVA, while the qualitative data was subjected to thematic analysis.

DETAILED DESCRIPTION:
Details of the Workshop Designing and facilitation: Faculty mentoring workshop with the title "Faculty Mentoring; building stronger by digging deeper" was designed as a two-day workshop of three hours each for the faculty members of the two institutions at separate times.

Workshop learning outcomes and activities: The learning outcomes of the workshop day 1 were, importance and benefits of faculty mentoring program, roles and responsibilities of mentors and mentees, the ethics and stages of any mentoring relationship. The activities used were group discussions and ethical dilemmas were demonstrated by role plays by the participants in groups of three. Day 2 agenda was developing a mentor or a mentee portfolio with special focus on self. The activities were personal Strength, Weakness, Opportunities and Threats (SWOT) analysis, goal setting for a mentor and a mentee and developing an action plan. Most of the day was dedicated to hands-on individual activities followed by voluntary sharing of the personal development goals and a discussion on the correct ways of framing goals and realistic ways of writing an actionable plan with milestones defining success.

Data Collection

Data Sources:

* Qualitative Data:

  * During Workshop: SWOT analysis, goals set and the action plan developed by each participant during the group activities and the individual hands-on sessions the workshop
  * Post workshop: Reflections of participants were requested to write the three things that they learnt, followed by the questions still in their mind and one change that they will make after the workshop
* Quantitative data

  * Pre workshop: The data of the faculty was collected before the workshop in terms of their title and years of experience.
  * Post workshop: feedback on the workshop's effectiveness was acquired by a questionnaire which was developed by department of Continuous Medical Education at Aga Khan University (Appendix A). The content, construct and criterion validity were checked before pilot testing by subject matter experts and it was ensured that questions were relevant to the objectives of the activity and was clear and understandable to the respondents. Responses were further categorized into levels of satisfaction: "Unsatisfactory," "Satisfactory," and "Excellent." Qualitative feedback was in alignment with the discussions during the workshop, with special focus on possible change in their mentoring practices after attending the workshop.

ELIGIBILITY:
Inclusion Criteria:

* Faculty members working full time in the medical college

Exclusion Criteria:

* The faculty not giving consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Personal Development Plan | At the end of the workshop (Day 2)
  Developing a personal development plan through SWOT analysis of self. The plan will identify the areas of mentoring that need improvement with the identified milestones and timelines

CONTACTS AND LOCATIONS:
Overall Officials: Saima Chaudhry, PhD, Study Chair — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan